CLINICAL TRIAL: NCT02094469
Title: A Multicenter, One Group, Open-label Study to Evaluate the Safety and Efficacy of Pletaal(Cilostazol) as BID for up to 24 Weeks Exposure in Subjects With Vasospastic Angina (STELLA Extension)
Brief Title: Safety and Efficacy Study of Cilostazol to Treat Vasospastic Angina
Acronym: STELLA_Ext
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 021-KOA-1302i
Record Dates: First submitted 2014-03-20; First posted 2014-03-21 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Vasospastic Angina
Keywords: Treatment for vasospastic angina
MeSH Terms: conditions — Angina Pectoris, Variant | interventions — Cilostazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cilostazol (Other): Cilostazol 50mg and 100mg
  Interventions: Drug: Cilostazol

INTERVENTIONS:
Drug: Cilostazol — Oral, Bid, 24 weeks
  Other Names: Pletaal

SUMMARY:
This study will be conducted in accordance with the local regulation of New Drug Application. Overall duration of this trial will be 3 years after approval of MFDS.

Each subject will participate around 26 weeks, which include the 24 weeks treatment period and 2 weeks safety follow up period. Withdrawn subjects due to efficacy after 4 weeks treatment will participate in 6 weeks in total including 2 weeks safety follow up. Withdrawn subjects with other reason also have 2 weeks follow up period.

DETAILED DESCRIPTION:
A Multicenter, One group, Open-label Study. Cilostazol will be treated for additional 24 weeks to the subject who had completed 021-KOA-1301i study. PletaalÒ(Cilostazol) is taken 100mg oral tablets bid during 2 3weeks after dosing of PletaalÒ(Cilostazol) 50mg oral tablets bid during 1 week. The dose can be adjusted by investigator's discretion during the study and the detailed method is described in the Protocol. Subject who has 2 or more chest pain at 4th week will be withdrawn from the study (But, subjects who show 50% or more of chest pain decrease compared to 1st week would not be withdrawn.). Subjects who participated in this trial will have 2 weeks follow-up after study completion.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 20 to 80 years, and subjects whose age at the time of enrollment was 80 in 021-KOA-1301i clinical trial and is 81 in this clinical trial
2. Subjects who completed 021-KOA-1301i clinical trial
3. Women of childbearing potential with negative pregnancy test at enrollment and who agree to practice a contraceptive measure throughout the clinical trial (e.g., hormonal contraceptives, intrauterine devices, condom + spermicidal agents, diaphragm + spermicidal agents, and partner's infertility)
4. Subjects who signed a written agreement indicating that they were given full explanations of the clinical trial and are willing to participate in the clinical trial

Exclusion Criteria:

1. Subjects who fell under one of the exclusion criteria at the time of enrollment for 021-KOA-1301i
2. Subjects who reported any of the following events, which fall under the exclusion criteria for KOA-1301i, between the initiation of 021-KOA-1301i participation and enrollment visit for 021-KOA-1302i

   * Myocardial infarction or myocardial infarction induced by vasospastic angina
   * Life-threatening vasospastic episodes (e.g., ventricular tachycardia, ventricular fibrillation, or syncope)
   * Stroke, intracranial hemorrhage, or transient ischemic attack (TIA)
   * Hemorrhage (hemophilia, capillary fragility, intracranial hemorrhage, upper gastrointestinal bleeding, urinary tract bleeding, hemoptysis, vitreous hemorrhage, etc.)
3. Subjects who are currently using any of the medications contraindicated in 021-KOA-1301i (excluding the investigational product of 021-KOA-1301i) at baseline
4. Subjects who meet the following criteria for baseline laboratory findings

   * severe anemia with hemoglobin ≤6.5 g/dl at baseline
   * Creatinine level ≥ 1.5 mg/dL at baseline
   * AST or ALT >3x ULN at baseline
   * Platelet count < 100,000mm3 at baseline
5. Pulse rate exceeding 100 bpm when measured for vital signs at baseline: Tachycardia
6. Hypotension with systolic pressure < 90mmHg at baseline
7. Uncontrolled hypertension defined as systolic pressure ≥ 160 mmHg or diastolic pressure ≥ 100 mmHg at baseline
8. QT prolongation defined as QTcB > 450 msec for men and QTcB > 470 msec for women at baseline
9. Women of childbearing potential with positive pregnancy test at baseline
10. Women who do not agree to practice a contraceptive measure, or are pregnant or lactating
11. Subjects who are not expected to have the potential to benefit from additional administration of Cilostazol, according to the investigator's judgment
12. Subjects otherwise judged by the investigator to be inappropriate for inclusion in the trial

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Proportion of the subjects whose chest pain was not present in the final 1 week/2 weeks after the 24-week treatment period | 24 weeks
  Proportion of the subjects whose chest pain was not present in the final 1 week/2 weeks after the 24-week treatment period

SECONDARY OUTCOMES:
secondary 1 | 24 week
  Change/rate of change in the frequency of chest pain in the final 1week/2 weeks after the 24-week treatment period compared to those in the final 1 week/2weeks of Amlodipine run-in period in 021-KOA-1301i
secondary 2 | 4 weeks
  Mean change in the intensity of chest pain in the final 1 week/2 weeks after the 24-week treatment period compared to that in the final 1 week/2weeks of Amlodipine run-in period in 021-KOA-1301i
secondary 3 | 4 weeks
  4-week cumulative rate of subjects withdrawn due to lack of efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Junghong Kim, MD, Principal Investigator — Yangsan Busan University Hospital
Locations (1):
- Yangsan Busan University Hospital, Busan, South Korea